CLINICAL TRIAL: NCT04888741
Title: A Multi-centre Phase II Trial of GVHD Prophylaxis Following Unrelated Donor Stem Cell Transplantation Comparing Thymoglobulin vs. Calcineurin Inhibitor or Sirolimus-based Post-transplant Cyclophosphamide
Brief Title: Methods of T Cell Depletion Trial (MoTD)
Acronym: MoTD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Birmingham (Other)
Collaborators: IMPACT (funded by NHS Blood & Transplant, Anthony Nolan and Leukaemia UK) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RG_19-116
Record Dates: First submitted 2021-03-03; First posted 2021-05-17 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Chronic Myelomonocytic Leukemia; Myelodysplastic Syndromes; Non Hodgkin Lymphoma; Hodgkin Lymphoma; Multiple Myeloma; Chronic Myelogenous Leukemia; Myelofibrosis
Keywords: GvHD; Allogeneic Stem Cell Transplant; AML; MDS; CML; CMML; NHL; HL; Cyclophosphamide; Thymoglobulin; Cyclosporin; Sirolimus; Mycophenolate Mofetil
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin; Hodgkin Disease; Multiple Myeloma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Primary Myelofibrosis | interventions — thymoglobulin; Cyclophosphamide; Cyclosporine; Sirolimus; Mycophenolic Acid

STUDY DESIGN:
Intervention Model Description: Patients eligible for entry into the trial will be randomised on a 1:1:1 ratio to receive either one of the experimental treatment arms or the control arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Arm Thymoglobulin + Cyclosporine + MMF (Active Comparator): Thymoglobulin is given as an intravenous infusion of 2.5 mg/kg/day over 2 days (days -2 and -1; total dose 5 mg/kg) via a central line through a 0.2 micron inline filter. Each dose will be infused over 6-8 hours. No test dose will be given. 30 minutes before Thymoglobulin, the patient should receive methylprednisolone 1mg/kg intravenously, 1g paracetamol PO and 10mg chlorphenamine IV. Patients should be monitored carefully and receive appropriate therapy for any infusion-related or anaphylactic reactions as per local policy.
  Patients will receive IV/PO cyclosporine according to local policy to begin on day -1 maintaining a trough level of 100-200 µg/L until day 90 before a subsequent taper in the absence of any active GvHD.
  MMF will be given IV/PO according to local policy at a dose of 1g TDS to begin on day -1 and discontinued on day 35 without taper if there is no evidence of active GvHD. In adults weighing <55kg, MMF should be given at a lower dose of 0.75g IV/PO TDS.
  Interventions: Drug: Thymoglobulin; Drug: Cyclosporine; Drug: Mycophenolate Mofetil
- Experimental arm (PTCy + Cyclosporine + MMF) (Experimental): Cyclophosphamide is given as an IV infusion of 50 mg/kg/day over 2 days (days 3 and 4; total dose 100 mg/kg) together with IV hydration and Mesna, as per local policy.
  Patients will receive IV/PO cyclosporine according to local policy to begin on day 5 maintaining a trough level of 100-200 µg/L until day 90 before a subsequent taper in the absence of active GvHD.
  MMF will be given IV/PO according to local policy at a dose of 1g TDS to begin on day 5 and discontinued on day 35 without taper if there is no evidence of active GvHD. In adults weighing <55kg, MMF should be given at a lower dose of 0.75g IV/PO TDS.
  Interventions: Drug: Cyclophosphamide; Drug: Cyclosporine; Drug: Mycophenolate Mofetil
- Experimental arm (PTCy + Sirolimus + MMF) (Experimental): Cyclophosphamide is given as an IV infusion of 50 mg/kg/day over 2 days (days 3 and 4; total dose 100 mg/kg) together with IV hydration and Mesna, as per local policy.
  Sirolimus will be initially given PO as a loading dose of 6 mg on day 5 followed by 2 mg daily; doses will be adjusted to maintain a trough level (in whole blood) of 8 to 14 ng/mL until day 60, thereafter 5-8 ng/mL until day 90. In the absence of active GvHD, the dose of sirolimus will be tapered from day 90. We recommend that the daily maintenance dose of sirolimus is reduced empirically to 0.5-1mg daily with concomitant treatment with a triazole anti-fungal agent.
  MMF will be given IV/O according to local policy at a dose of 1g TDS to begin on day 5 and discontinued on day 35 without taper if there is no evidence of active GvHD. In adults weighing <55kg, MMF should be given at a lower dose of 0.75g IV/PO TDS.
  Interventions: Drug: Cyclophosphamide; Drug: Sirolimus; Drug: Mycophenolate Mofetil

INTERVENTIONS:
Drug: Thymoglobulin — GVHD prophylaxis
  Other Names: ATG
  Arms: Control Arm Thymoglobulin + Cyclosporine + MMF
Drug: Cyclophosphamide — Post transplant cyclophosphamide strategy for GVHD prophylaxis
  Arms: Experimental arm (PTCy + Cyclosporine + MMF); Experimental arm (PTCy + Sirolimus + MMF)
Drug: Cyclosporine — immunosuppressant
  Arms: Control Arm Thymoglobulin + Cyclosporine + MMF; Experimental arm (PTCy + Cyclosporine + MMF)
Drug: Sirolimus — immunosuppressant
  Arms: Experimental arm (PTCy + Sirolimus + MMF)
Drug: Mycophenolate Mofetil — immunosuppressant
  Other Names: MMF

SUMMARY:
A multi-centre phase II trial of GvHD prophylaxis following unrelated donor stem cell transplantation comparing Thymoglobulin vs. Calcineurin inhibitor or Sirolimus-based post-transplant cyclophosphamide.

DETAILED DESCRIPTION:
This is a prospective, phase II, adaptive, multicentre, randomised clinical trial in patients undergoing reduced intensity conditioned (RIC) unrelated donor allogeneic stem cell transplantation (allo-SCT). The trial will compare the novel graft-versus-host disease (GvHD) prophylaxis regimens of post-transplant cyclophosphamide (PTCy) + Calcineurin inhibitor (CNI) (PTCy-CNI) or PTCy + Sirolimus to a current standard-of-care involving the use of T-cell depletion with Thymoglobulin. Patients will be minimised at randomisation by their randomising centre, disease risk score (low/intermediate or high/very high) and human leukocyte antigen (HLA) match (10/10 or 9/10). Patients eligible for entry into the trial will be randomised on a 1:1:1 ratio to receive either one of the experimental treatment arms or the control arm.

The primary objective is to compare GvHD-free, relapse-free Survival (GRFS) in patients treated with the GvHD prophylaxis regimens PTCy-CNI, PTCy-Sirolimus or T-cell depletion with Thymoglobulin.

The secondary objectives are to evaluate the cumulative incidence of acute GvHD (aGvHD), the cumulative incidence of moderate and severe chronic GvHD (cGvHD), the cumulative incidence of non-relapse mortality (NRM), overall survival (OS), progression-free survival (PFS), immune suppression-free survival, the cumulative incidence of engraftment, the incidence of full donor chimerism, the cumulative incidence of infection requiring inpatient admission, the number of inpatient days, the timing and dose of donor lymphocyte infusion (DLI), the cumulative incidence of Epstein-Barr virus (EBV) related-post transplant lymphoproliferative disease (PTLD), the number of doses rituximab administered for EBV reactivation, quality of life (QoL), the cumulative incidence of haemorrhagic cystitis, the cumulative incidence of cytomegalovirus (CMV) viraemia and CMV end-organ disease and safety and tolerability.

The scientific research will address the questions about how plasma biomarkers for GvHD predict GvHD and non-relapse mortality following T-cell depleted methods of transplantation and how the different methods of T-cell depletion impact on immune function and re-constitution.

Outcome Measures

Primary Outcome Measure:

• GvHD-free, relapse-free survival at 1 year

Secondary Outcome Measures:

* Cumulative incidence of acute grade II-IV and III-IV GvHD at 1 year
* Cumulative incidence of moderate and severe chronic GvHD at 1 year
* Cumulative incidence of NRM at 1 year
* Overall survival at 1 year
* Progression-free survival at 1 year
* Immune suppression-free survival at 1 year
* Cumulative incidence of engraftment at 1 year
* The incidence of full donor chimerism at 100 days
* The cumulative incidence of infection requiring inpatient admission at 1 year
* The number of inpatient days during first 12 months
* The timing and dose of DLI for mixed chimerism, persistent disease or relapse
* Cumulative incidence of EBV-related PTLD
* The number of doses of rituximab administered for EBV reactivation during first 12 months
* QoL measured by FACT-BMT questionnaire at baseline, 6 months and 12 months
* Cumulative incidence of patients with haemorrhagic cystitis at 1 year
* Cumulative incidence of CMV viremia and CMV end-organ disease at 1 year
* Safety defined as the incidence of ≥ grade 3 toxicities reported as per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.0
* Tolerability defined to be the number of patients able to complete therapy as scheduled

Exploratory Outcome Measures:

The scientific research will address the following questions:

1. Do plasma biomarkers for GvHD predict GvHD and non-relapse mortality following T-cell depleted methods of transplantation?
2. Do PTCy methods increase T cell receptor repertoire diversity (as measured by TCR DNA sequencing) compared to ATG-based T cell depletion?
3. How do the different methods of T-cell depletion impact upon donor Treg reconstitution?
4. How do the different methods of T-cell depletion impact upon thymic function as evaluated by measurement of recent thymic emigrants?
5. Are PTCy methods of TCD associated with better preservation of virus-specific immunity (as measured by tetramer or ex vivo functional immune responses)?

Patient Population

Adults considered suitable for an allo-SCT with the following haematological malignancies will be recruited to this trial:

* Acute Myeloid Leukaemia (AML)
* Acute lymphoblastic leukaemia (ALL)
* Chronic myelomonocytic leukemia (CMML)
* Myelodysplastic syndromes (MDS)
* Non-Hodgkin lymphoma (NHL)
* Hodgkin lymphoma (HL)
* Multiple myeloma (MM)
* Chronic lymphocytic leukaemia (CLL)
* Chronic myeloid leukaemia (CML)
* Myelofibrosis

Sample Size:

Up to 400 patients will be randomised to the MoTD trial across IMPACT centres.

Trial Duration:

Patients will be recruited over 48 months. Patients will be followed up for a minimum of 1 year.

MoTD Trials Office Contact Details:

MoTD trials office, Centre for Clinical Haematology, Queen Elizabeth Hospital, Edgbaston, Birmingham, B15 2TH Tel: 0121 371 7858 Email: MoTD@trials.bham.ac.uk

ELIGIBILITY:
Inclusion Criteria:

* Availability of suitably matched unrelated donor (9/10 or 10/10)
* Planned to receive one of the following RIC protocols:

  * Fludarabine-Melphalan (Fludarabine 120-180mg/m2 IV; melphalan ≤ 150mg/m2 IV)
  * BEAM or LEAM (carmustine 300mg/m2 IV or lomustine 200mg/m2 IV with: etoposide 800 mg/m2 IV; cytarabine 1600mg/m2 IV; melphalan 140mg/m2 IV)
  * Fludarabine-Busulphan (Fludarabine 120-180mg/m2 IV; Busulphan ≤ 8mg/kg PO or 6.4mg/kg IV)
  * Fludarabine- Treosulfan (Fludarabine 150mg/m2 IV; Treosulfan 30g/m2 IV)
* Planned use of PBSCs for transplantation
* Planned allo-SCT for one of the following haematological malignancies:

  * AML in CR (patients enrolled onto the COSI trial are not eligible for this study)
  * ALL in CR (patients enrolled onto the ALL-RIC trial are not eligible for this study)
  * CMML <10% blasts
  * MDS <10% blasts (patients enrolled onto the COSI trial are not eligible for this study)
  * NHL in CR/PR
  * HL in CR/PR
  * MM in CR/PR
  * CLL in CR/PR
  * CML in 1st or 2nd chronic phase
  * Myelofibrosis
* Age 16-70 years
* Females of and male patients of reproductive potential (i.e., not post-menopausal or surgically sterilised) must agree to use appropriate, highly effective, contraception from the point of commencing therapy until 12 months after transplant

Exclusion Criteria:

* Use of any method of graft manipulation (excluding storage of future DLI)
* Use of alemtuzumab or any method of T cell depletion except those that are protocol-defined
* Known hypersensitivity to study drugs or history of hypersensitivity to rabbits
* Pregnant or lactating women
* Adults of reproductive potential not willing to use appropriate, highly effective, contraception during the specified period
* Life expectancy <8 weeks
* Active HBV or HCV infection
* Organ dysfunction defined as:

  * LVEF <45%
  * GFR <50ml/min
  * Bilirubin >50µmol/l
  * AST/ALT>3 x ULN
* Participation in COSI or ALL-RIC trials
* Contraindication to treatment with the study drugs (Thymoglobulin, cyclophosphamide, sirolimus, ciclosporin and mycophenolate mofetil) as detailed in each study drug SPC.
* Patient has any other systemic dysfunction (e.g., gastrointestinal, renal, respiratory, cardiovascular) or significant disorder which, in the opinion of the investigator would jeopardise the safety of the patient by taking part in the trial.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-02-22 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
GVHD-free, relapse-free survival | at 1 year
  GVHD assessment scoring will be performed as per the modified Glucksberg criteria (revised by MAGIC) and the National Institutes of Health (NIH) criteria. GvHD-free, relapse-free survival (GRFS) defined as the time from date of day 0 (defined as the day of stem cell infusion) to the date of first event or death from any cause. An event is defined as GvHD (both acute and chronic), relapse or progression. Patients who are alive and event free at the end of the trial will be censored at their date of last follow-up

SECONDARY OUTCOMES:
Cumulative incidence of acute grade II-IV and III-IV GvHD | at 1 year
  GVHD assessment scoring will be performed as per the modified Glucksberg criteria (revised by MAGIC) and the National Institutes of Health (NIH) criteria. GvHD-free
Cumulative incidence of moderate and severe chronic GvHD | at 1 year
  GVHD assessment scoring will be performed as per the modified Glucksberg criteria (revised by MAGIC) and the National Institutes of Health (NIH) criteria. GvHD-free
Cumulative incidence of NRM | at 1 year
  Non-relapse mortality (NRM) is defined as the time from day 0 to date of non-relapse death. Patients who die post-relapse from any other cause will be considered a competing risk and patients alive at the end of the trial will be censored at their date last seen.
Overall survival | at 1 year
  Overall survival (OS) is defined as the time from day 0 to date of death, from any cause. Patients who are alive at the end of the trial will be censored at their date last seen.
Progression-free survival | at 1 year
  Progression-free survival (PFS) is defined as the time from day 0 to date of first relapse/progression or death from any cause. Patients who are alive and progression free at the end of the trial will be censored at their date last seen.
Immune suppression-free survival | at 1 year
  Immune suppression-free survival is defined as time from day 0 to the date of first immunosuppressive agent use. Patients who are alive and immune suppression free at the end of the trial will be censored at their date last seen
Cumulative incidence of engraftment | at 1 year
  Cumulative incidence of engraftment defined as time from day 0 to date of engraftment (Neutrophil engraftment defined to be the first of 3 consecutive days a neutrophil count ≥ 0.5×〖10〗^9/L is reached and platelet engraftment defined to be the first of 3 consecutive days an unsupported platelet count ≥ 20×〖10〗^9/L is reached). Patients who relapse/progress or die prior to relapse, progression or engraftment will be considered a competing risk at their date of relapse/progression for the former and date of death for the latter. Patients alive and engraftment free at the end of the trial will be censored at their date last seen.
The incidence of full donor chimerism | at 100 days
  Engraftment will be assessed by lineage specific chimerism measurements. Lineage specific chimerism in both whole blood and T-cell compartments (where possible) will be assessed as per local procedure, performed at 3 monthly intervals for the first 12 months post-transplant; at day 100 and then months 6, 9 and 12. Tests should be performed in local laboratories.
The cumulative incidence of infection requiring inpatient admission | at 1 year
  The cumulative incidence of infection requiring inpatient admission measured by blood test and tissue culture at 1 year
The number of inpatient days | during first 12 months
  The sum of inpatients days
The timing of mixed chimerism, persistent disease or relapse | during first 12 months
  We will be recording the time (days, post-transplant) whenever mixed chimerism, persistent disease or relapse occurred post transplant
Cumulative incidence of EBV-related PTLD | during first 12 months
  Measured by blood sample, EBV PCR testing.
The number of doses of Rituximab administered for EBV reactivation | during first 12 months
  We will collect the number of doses every time the patient will receive Rituximab whenever there is EBV reactivation
QoL measured by FACT-BMT questionnaire | at baseline, 6 months and 12 months
  QoL measured by FACT-BMT questionnaire at baseline, 6 months and 12 months. FACT-BMT Questionnaire uses Units on a scale 0-4, higher scores mean a better outcome.
Cumulative incidence of patients with haemorrhagic cystitis | at 1 year
  Cumulative incidence of patients with haemorrhagic cystitis measured by blood and urine sample at 1 year
Cumulative incidence of CMV viremia and CMV end-organ disease | at 1 year
  Cumulative incidence of CMV viremia and CMV end-organ disease measured by blood sample at 1 year
Safety defined as the incidence of ≥ grade 3 toxicities reported as per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) V4.0 | from the date of commencement of protocol defined treatment until 28 days after the administration of the last dose of IMP.
  . Safety defined as the incidence of ≥ grade 3 toxicities reported as per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.0. Details of all AEs will be documented and reported from the date of commencement of protocol defined treatment until 28 days after the administration of the last dose of IMP. Serious AEs will be reported from the date of consent.
Tolerability defined to be the number of patients able to complete therapy as scheduled | during first 12 months
  Tolerability defined to be the number of patients able to complete therapy as scheduled (excluding any patients who discontinued treatment due to toxicities
Dose of Donor lymphocyte infusion (DLI) for mixed chimerism, persistent disease or relapse | during first 12 months
  We will be collecting the dose of DLI (CD3 Cells/kg) whenever required for mixed chimerism, persistent disease or relapse

CONTACTS AND LOCATIONS:
Overall Officials: Ronjon Professor Chakraverty, Study Director — Oxford Cancer & Haematology Centre, The Churchill Hospital, Old Road - Headington, Oxford, OX3 7LE Email: ronjon.chakraverty@ndcls.ox.ac.uk
Locations (15):
- United Kingdom (15):
  - University Hospital of Wales, Cardiff, Wales
  - Queen Elizabeth Hospital, Birmingham
  - Bristol Haematology and Oncology Centre, Bristol
  - Addenbrookes Hospital, Cambridge
  - Queen Elizabeth Hospital Glasgow, Glasgow
  - St Jame's University Hospital, Leeds
  - University College London Hospital, London
  - King's College Hospital, London
  - Hammersmith Hospital, London
  - Manchester Royal Infirmary, Manchester
  - The Christie, Manchester
  - Freeman Hospital, Newcastle upon Tyne
  - Nottingham City Hospital, Nottingham
  - Churchill Hospital, Oxford
  - Derriford Hospital, Plymouth

IPD SHARING:
Plan to Share IPD: No